CLINICAL TRIAL: NCT05816252
Title: A Phase II Study of SKB264 as Monotherapy or as Combination Therapy in Subjects With Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of SKB264 (MK-2870; Sac-TMT) for the Treatment of Participants With Advanced or Metastatic Non-small Cell Lung Cancer (SKB264-II-04) (MK-2870-003)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Klus Pharma Inc. (Industry)
Collaborators: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-II-04; MK-2870-003 (Other: Merck Sharp & Dohme LLC); 2023-507270-41-00 (EU CTIS Number)
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Injections; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 1L NSCLC, EGFR/ALK negative and PD-L1 TPS ≥ 1% (Experimental): SKB264 (Dose Level 1) + Pembrolizumab
  Interventions: Drug: SKB264; Drug: Pembrolizumab
- Cohort 3 1L NSCLC, EGFR/ALK negative, regardless of PD-L1 expression level (Experimental): SKB264 (Dose Level 1') + Pembrolizumab + Carboplatin
  Interventions: Drug: SKB264; Drug: Pembrolizumab; Drug: Carboplatin
- Cohort 4 1L NSCLC, EGFR/ALK negative, regardless of PD-L1 expression level (Experimental): SKB264 (Dose Level 1'') + Pembrolizumab + Carboplatin
  Interventions: Drug: SKB264; Drug: Pembrolizumab; Drug: Carboplatin
- Cohort 5 NSCLC with EGFR mutation and after failure of EGFR TKI therapy (Experimental): SKB264 (Dose Level 1') + Carboplatin
  Interventions: Drug: SKB264; Drug: Carboplatin
- Cohort 6 NSCLC with EGFR mutation and after failure of EGFR TKI therapy (Experimental): SKB264 (Dose Level 1'') + Carboplatin
  Interventions: Drug: SKB264; Drug: Carboplatin
- Cohort 7 1L NSCLC with EGFR mutation (Experimental): SKB264 (Dose Level 1) + Osimertinib
  Interventions: Drug: SKB264; Drug: Osimertinib
- Cohort 7-1 1L NSCLC with EGFR mutation (Experimental): SKB264 (Dose Level 2) + Osimertinib
  Interventions: Drug: SKB264; Drug: Osimertinib
- Cohort 9 2/3L NSCLC EGFR/ALK negative (Experimental): SKB264 (Dose Level 1)
  Interventions: Drug: SKB264

INTERVENTIONS:
Drug: SKB264 — intravenous (IV) infusion (Q2W or Q3W)
  Other Names: MK-2870; Sacituzumab Tirumotecan (Sac-TMT)
Drug: Pembrolizumab — intravenous (IV) infusion (400mg, Q6W)
  Other Names: MK-3475
  Arms: Cohort 1 1L NSCLC, EGFR/ALK negative and PD-L1 TPS ≥ 1%; Cohort 3 1L NSCLC, EGFR/ALK negative, regardless of PD-L1 expression level; Cohort 4 1L NSCLC, EGFR/ALK negative, regardless of PD-L1 expression level
Drug: Carboplatin — intravenous (IV) infusion (AUC5, Q3W)
  Other Names: Carboplatin for injection
  Arms: Cohort 3 1L NSCLC, EGFR/ALK negative, regardless of PD-L1 expression level; Cohort 4 1L NSCLC, EGFR/ALK negative, regardless of PD-L1 expression level; Cohort 5 NSCLC with EGFR mutation and after failure of EGFR TKI therapy; Cohort 6 NSCLC with EGFR mutation and after failure of EGFR TKI therapy
Drug: Osimertinib — 80mg, QD
  Other Names: Osimertinib Mesylate
  Arms: Cohort 7 1L NSCLC with EGFR mutation; Cohort 7-1 1L NSCLC with EGFR mutation

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and objective response rate of SKB264 as combination with therapy in subjects with advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label study of SKB264 as combination therapy or monotherapy in subjects with NSCLC. Approximately 498 subjects will be enrolled in this study including around 88 subjects for the safety run-in period and 410 subjects for the expansion period.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be at least 18 years of age on day of signing informed consent, regardless of gender;
2. Subjects with histologically or cytologically confirmed locally advanced or metastatic NSCLC ;
3. Subjects for NSCLC should be confirmed to be EGFR (Epidermal growth factor receptor) wild-type and ALK (Anaplastic lymphoma kinase) fusion gene negative; or confirmed to harbor EGFR mutation;
4. Locally advanced or metastatic NSCLC subjects without actionable EGFR mutations and ALK fusion genes, no prior systemic treatment; subjects with EGFR mutation, no prior systemic treatment or failed prior EGFR-TKI (Tyrosine kinase inhibitor) treatment;
5. Subjects are able to provide tumor blocks or slides before the first dose of study intervention;
6. Subject must have at least one radiographically measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria;
7. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1;
8. Life expectancy at least 3 months for the subject;
9. Adequate organ function;
10. Subjects must have recovered from all toxicities led by prior treatment;
11. Contraceptive methods used by male and female subjects must comply with contraceptive methods of local regulations for clinical study subjects;
12. Subjects should voluntarily participate in the study, sign the ICF, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria

1. Subjects with mixed SCLC histopathological features;
2. Subjects with a known history of prior malignancy;
3. Subjects with known meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, or active central nervous system (CNS) metastases;
4. Subjects with ≥ Grade 2 peripheral neuropathy;
5. Subjects who had arteriovenous thromboembolic events, tumor invasion/encasement of vital organs/vessels, risk of esophageal-tracheal/pleural fistula, or current superior vena cava syndrome;
6. Subjects with active inflammatory bowel disease or previous clear history of inflammatory bowel disease;
7. Subjects who suffer from cardiovascular diseases of clinical significance;
8. Subjects with a history of interstitial lung disease (ILD)/non-infectious pneumonitis that required steroids;
9. Subjects with uncontrolled systemic disease as judged by the Investigator;
10. Subjects with active autoimmune disease that required systemic treatment in the past 2 years;
11. Subjects with active hepatitis B or hepatitis C;
12. Subjects with known history of Human Immunodeficiency Virus (HIV)
13. Subjects with known active tuberculosis;
14. Subjects with known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study;
16. Subjects whose condition deteriorated rapidly, such as severe changes in performance status, during the screening process prior to the first dose of study intervention;
17. Subjects with other circumstances that, in the opinion of the Investigator, are not appropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From subject sign the informed consent form (ICF) to 30 days after the last dose of study treatment, up to approximately 36 months
  Dose-limiting toxicity (DLT); Incidence and severity of adverse events (AEs); Discontinuation of study treatment due to AEs
ORR | The proportion of subjects with a confirmed complete response (CR) or partial response (PR), up to approximately 36 months
  Objective response rate (ORR) per RECIST v1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | From baseline until disease progression, death, or other protocol defined reason, up to approximately 36 months
  For subjects with a confirmed CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until radiographic disease progression or death due to any cause, whichever occurs first
Progression-free survival (PFS) | From baseline until disease progression, death, or other protocol defined reason, up to approximately 36 months
  The time from first dose of study intervention to first documentation of radiographic disease progression or death due to any cause, whichever occurs first
Overall survival (OS) | From baseline until death due to any cause, up to approximately 36 months
  the time period from the start of study intervention to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (50):
- China (27):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital (Chongqing Cancer Hospital), Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yatsen University Cancer Center Huangpu Hos, Guangzhou, Guangdong
  - Guangxi Cancer Hospital/ Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University(Heyi Compus), Zhengzhou, Henan
  - Henan Cancer Hospital,Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Chinese Medical University(Heping Compus), Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Georgia (3):
  - ISR-GEO Med Res Clin Healthycore, Tbilisi
  - LLC "Todua Clinic", Tbilisi
  - Ltd New Hospitals, Tbilisi
- Romania (2):
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca, Cluj
  - Centrul de Oncologie Sf. Nectarie, Craiova, Dolj
- South Korea (5):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Inje University Haeundae Paik Hospital, Busan
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (8):
  - Hospital Universitario Puerta De Hierro De Majadahonda, Majadahonda, Madrid
  - Hospital Universitario QuirónSalud Madrid, Pozuelo de Alarcón, Madrid
  - Micancer Center S.L.P., Barcelona
  - Hospital Universitari Dexeus Grupo Quironsalud, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clinico Universitario De Valencia, Valencia
- Turkey (Türkiye) (5):
  - Medical Park Seyhan Hospital, Adana
  - Adana City Training and Research Hospital, Adana
  - Gulhane Egitim ve Arastirma Hastanesi Tibbi Onkoloji Klinigi, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara